CLINICAL TRIAL: NCT02747420
Title: Randomized Controlled Trial of PTNS Versus Sham Efficacy in Treatment of Bladder Pain Syndrome
Brief Title: PTNS Versus Sham Efficacy in Treatment of BPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01447
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Interstitial Cystitis Bladder Pain Syndromes
Keywords: Posterior Tibial Nerve Stimulation, Bladder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Post Tibial Nerve Stimulation Group (PTNS) (Experimental)
  Interventions: Device: NURO TM
- Sham Group (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: NURO TM — The lower extremity will be palpated and a needle insertion site will be identified 5 cm from the medial malleolus and posterior to the tibia. Between the posterior margin of the tibia and the soleus muscle, a 34-gauge acupuncture-like needle will be inserted 3-4 cm to the tibial nerve. A grounding pad will be placed on the bottom of the foot just below the smallest toe. An inactive grounding pad will be placed on top of the foot above the small toe to be consistent with the sham pad placement. The needle and grounding pad will be connected to the stimulator and the stimulation will be increased from 0 to 10 Milli-ampere. The needle will be taped. The electrical current will be set by the subject and the mA will be recorded. A 30 minute stimulation session will be given at 20 Hz.
  Other Names: Neuromodulation system, Medtronic Device Model # 3533; stimulator model NURO 100
  Arms: Post Tibial Nerve Stimulation Group (PTNS)
Device: Sham — A needle will be inserted into the lower extremity approximately 5 cm cephalad from the medial malleolus and posterior to the tibia. A sham needle will be used a the tibial nerve insertion site. This will stimulate needle placement without puncturing the skin. The needle will be taped in place. The "grounding pad" from the transcutaneous electrical nerve stimulation (TENS) unit device will be placed on the bottom of the foot below the smallest toe. Another electrode will be placed on the top of the foot above the small toe for conduction. The TENS electrode will be connected to the TENS unit, at 20 Hz (the same as the PTNS group). The unit will be turned on and the stimulation will be increased to the subject's first sensory level. The subject will sense stimulation to either the bottom of the foot or the toe. the TENS unit will be on for a 30 minute test period. The TENS unit will be removed and the needle will be discarded.
  Arms: Sham Group

SUMMARY:
This is a prospective, single center, double-blind, randomized, controlled trial comparing the efficacy of percutaneous tibial nerve stimulation to sham in the treatment of Bladder Pain Syndrome/Interstitial Cystitis (BPS/IC) through 12 weeks of therapy.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the efficacy of the systematic effects of posterior tibial nerve stimulation (PTNS) treatment compared to an inactive sham intervention in female subjects with interstitial cystitis/bladder pain syndrome (IC/BPS) in an intent-to-treat analysis. The primary outcome measure will be the Patient Global Impression of Improvement (PGI-I) a single item questionnaire assessing overall impression of improvement over time at the initial 12 weeks endpoint.

It is hypothesized that subjects randomized to the PTNS arm will demonstrate a greater improvement in both pain and quality of life scores, when compared with subjects who are randomized to the sham arm.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old with visual analog scale > 5
* Cessation of all analgesics or other medication for pain for at least 2 weeks prior to the PTNS intervention
* Discontinuation of any other electrical stimulation methods for 3 months prior to PTNS intervention.
* Capable of giving informed consent
* Ambulatory
* Capable and willing to follow all study-relation procedures

Exclusion Criteria:

* Patients pregnant or planning to become pregnant during the study duration
* Botox use in pelvic floor muscles within the last year
* Current urinary or vaginal infections
* Current use of Interstim device
* History of a cardiac pacemaker
* Diagnosis of neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01-18 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brucker, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post Tibial Nerve Stimulation Group (PTNS) | Sham Group
Started | 18 | 22
Completed | 11 | 18
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post Tibial Nerve Stimulation Group (PTNS) | Sham Group | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (18.3) | 51.7 (18.2) | 51.2 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Patient Global Impression of Improvement (PG-I) Score = 1 or 2
Description: A single item questionnaire assessing overall impression of improvement over time at the initial 12 weeks endpoint.
  Patients are asked to describe their condition compared to how it was before intervention on a scale from 1 to 7:
  Very much better = 1 Much better = 2 A little better = 3 No change = 4 A little worse = 5 Much worse = 6 Very much worse = 7
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Post Tibial Nerve Stimulation Group (PTNS) | Sham Group
Number analyzed (Participants) | 18 | 22
Participants | 2 | 4

2. Secondary Outcome: Visual Analog Scale (VAS)
Description: Quality of Life Scores
Time Frame: 12 Weeks
Reporting Status: Not Posted

3. Secondary Outcome: O'Leary-Sant Pain Scores
Description: pain intensity, location of pain and associated symptoms
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Over Active Bladder-Questionnaire (OAB-Q)
Description: This will allow for evaluation of subjects with concomitant overactive bladder and painful bladder syndrome characteristics.
Time Frame: 12 Weeks
Reporting Status: Not Posted

5. Secondary Outcome: The SF-12 (Short Form) Health Scale
Description: Used to evaluate quality of life of each subject at the three analysis intervals.
Time Frame: 12 Weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Post Tibial Nerve Stimulation Group (PTNS) | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT02747420/Prot_SAP_000.pdf